CLINICAL TRIAL: NCT00175591
Title: The Effect of Femoral Nerve Block on Opioid Requirements Following Femoral Fracture Fixation With Flexible Nails in the Paediatric Population: A Double Blind, Prospective Randomized Clinical Trial
Brief Title: The Effect of Femoral Nerve Block on Opioid Requirements After Surgery for a Femur Fracture in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H05-70077; W05-0025
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pain, Postoperative
Keywords: Femur fracture; morphine sparing; preemptive analgesia; Post-operative pain and post- operative opioid use
MeSH Terms: conditions — Pain, Postoperative; Femoral Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Administration of a femoral nerve block (bupivacaine HCL) — No details specified

SUMMARY:
This study evaluates the effect of a femoral nerve block on opioid requirements following femoral fracture fixation with flexible nails in the paediatric population. This is a double blind, prospective randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Femoral shaft fracture requiring intra-medullary nailing
* Surgery performed within 24 hours of injury
* Ability of child or family to use patient-controlled analgesia (PCA)
* No allergy or sensitivity to bupivacaine
* Informed consent and assent

Exclusion Criteria:

* Open femur fractures
* Closed fractures needing open reduction
* Fractures associated with neurovascular complications
* Fractures associated with compartment syndrome
* Repeat femoral surgeries
* Patients who received a femoral nerve block more than 1 hour prior to surgery
* Complex associated injuries or pre-existing condition that will delay time to ambulation
* Children who are allergic and/or sensitive to bupivacaine

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine requirement; the average 8 hour morphine requirement (mcg/kg/hr) will be recorded | until patient discharge

SECONDARY OUTCOMES:
Pain rating | immediately post-op
Sedation/pruritis/nausea/vomiting/urinary retention/respiratory rate | every 8 hours
Time to discharge | from end of surgery
Time (hours) from end of surgery to sitting on bed with legs hanging over the side

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada